CLINICAL TRIAL: NCT02967432
Title: Randomized Controlled Trial of Mupirocin to Reduce Staphylococcus Aureus Colonization in Infants Hospitalized in a Neonatal Intensive Care Unit
Brief Title: Mupirocin to Reduce Staphylococcus Aureus Colonization in Infants Hospitalized in a NICU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crouse Hospital (Other)
Collaborators: Jana Shaw, MD (Unknown); Steven Gross, MD (Unknown); David Martin, RN (Unknown); Dale Franz, RPh (Unknown); Rachel Carey (Unknown)
Responsible Party: Principal Investigator, Melissa Nelson, MD, Attending Physician, Neonatologist, Crouse Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Crouse Hospital 2016.0125
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Staphylococcus
Keywords: Staphylococcus aureus; Staphylococcal colonization; Staphylococcal infection; Mupirocin; Mupirocin-resistance
MeSH Terms: conditions — Staphylococcal Infections | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mupirocin (Experimental)
  Interventions: Drug: Mupirocin Topical Ointment
- Petroleum jelly (Placebo Comparator)
  Interventions: Drug: Petroleum Jelly

INTERVENTIONS:
Drug: Mupirocin Topical Ointment — Mupirocin ointment 1/2 inch ribbon applied topically to each nare and umbilicus twice daily for 5 days; repeat treatment courses possible.
  Arms: Mupirocin
Drug: Petroleum Jelly — Petroleum jelly ointment 1/2 inch ribbon applied topically to each nare and umbilicus twice daily for 5 days; repeat treatment courses possible.
  Arms: Petroleum jelly

SUMMARY:
The purpose of this study is to determine whether or not mupirocin treatment results in S. aureus decolonization in affected NICU patients.

DETAILED DESCRIPTION:
This randomized controlled trial of mupirocin treatment of MSSA- and MRSA-colonized infants aims to determine whether or not mupirocin treatment results in S. aureus decolonization in affected NICU patients. MSSA- or MRSA-colonized patients who enroll in the study will be randomized to either a treatment group (treatment with mupirocin) or control group (treatment with placebo). A combination of active surveillance and targeted decolonization will qualitatively and quantitatively enable assessment of any changes in S. aureus colonization in study patients. The primary outcome measure will be the number of MSSA/MRSA patient colonization days in the treatment versus control groups. Secondary outcome measures will include the proportion of persistently colonized patients at each subsequent weekly screening interval in the treatment versus control group, incidence and timing of MSSA/MRSA recolonization in the treatment group, incidence of invasive infections with S. aureus in the treatment versus control group, incidence of mupirocin-resistance in treatment versus control group, and incidence of MSSA/MRSA colonization after NICU discharge in the treatment versus control group.

STUDY PROCEDURES

Current standard of care in the NICU includes active universal screening of all admitted patients weekly for MSSA/MRSA colonization and contact precautions for MRSA-positive patients. No universal or targeted decolonization procedures are currently utilized. NICU patients who screen positive for MSSA/MRSA colonization will be approached for participation in this study and consent will be obtained from a parent within 2 days of the initial positive screening result by a neonatologist. At time of enrollment, patients will be randomized to either the treatment or control group. The pharmacy team will assign randomization; all NICU staff will be blinded to the patient's study group assignments throughout their admission. The treatment group will receive mupirocin ointment applied twice daily inside the nares and to the skin around the umbilicus for five days. The control group will receive a placebo ointment (petroleum jelly) applied in an identical fashion. The control group will not receive mupirocin ointment at any time, regardless of colonization status. If patients have recurrent positive MSSA/MRSA screens during the study, they may receive additional identical courses of treatment with either mupirocin or placebo based on their study group assignment.

The mupirocin and placebo petroleum jelly ointments will be supplied by the Crouse Hospital pharmacy and sent to the NICU daily for twice daily application by the nursing staff. Both groups will receive a ½ inch ribbon topical application of mupirocin or petroleum jelly ointment according to their assignment around the umbilicus and a ½ inch ribbon inside each nare. The neonatal nursing staff will receive appropriate education regarding the application technique and study protocol prior to study initiation. The cost of the mupirocin and placebo ointments will be paid for by Neonatal Associates of Central New York, LLC, and patients will not receive any fee for this service.

Colonization with MSSA/MRSA will be screened weekly on Mondays, in line with current Crouse Hospital NICU standard of care. MSSA/MRSA screening is performed by polymerase chain reaction (PCR). Sample collection involves swabbing an infant's nares, umbilicus, and groin with a cotton-tipped applicator. The swab tip is then sent to the Crouse Hospital Laboratory for Staphylococcus species identification. There will be no additional costs associated with these screenings, as this is already standard of care. Mupirocin resistance will be assessed by disk diffusion assay with E-test methodology to determine MICs. The costs associated with this additional test will be paid for by Neonatal Associates of Central New York, LLC, and patients will not receive any fee for this service. An additional MSSA/MRSA screen will be performed approximately 2 months after discharge at a patient's primary care physicians' office visit. Sample collection procedures will be identical to the screens performed at Crouse, and the screens will be sent to Laboratory Alliance of Central New York's Microbiology Department for testing. Results will be made available to the principal investigator. The costs associated with this additional outpatient screening test will be paid for by Neonatal Associates of Central New York, LLC, and patients will not receive any fee for this service.

Routine Crouse Hospital NICU policies regarding the use of contact precautions for any MRSA colonized infant will continue during the study period. If an infant enrolled in the study displays signs or symptoms concerning for infection, diagnostic evaluation and treatment will be guided by the attending neonatologist, not deviating from the current NICU standard of care. Parents are notified if their infant screens positive for MRSA colonization and if any diagnostic evaluation was performed on their infant. Current standards of infection prevention, such as aggressive and consistent hand hygiene, sterile procedure policies, etc. will be continued during this study.

Baseline patient demographics and clinical characteristics and outcomes will be collected on every study subject, including: birth weight, sex, gestational age, birth hospital, mode of delivery, maternal age, length of rupture of membranes, chorioamnionitis, documented maternal MRSA history when available, maternal antibiotic exposure, maternal drug abuse history, respiratory support throughout hospitalization, central line access, number of days on TPN, maternal breast milk and/or formula use, gavage feeding, surgery, grade III/IV intraventricular hemorrhage (IVH), necrotizing enterocolitis (NEC), spontaneous intestinal perforation (SIP), clinical condition and gestational age at time of any infectious evaluation, description of any positive infection (cerebrospinal fluid, blood, urine, pustule, abscess, osteomyelitis, endocarditis), antibiotic exposure (agent, antibiotic days), length of hospital stay, discharge disposition, and MSSA/MRSA colonization screening results.

The number of MSSA/MRSA patient colonization days will be determined and compared between the treatment and control groups. The proportion of persistently colonized, decolonized, and recolonized study subjects at each subsequent weekly screening interval in each study group will be determined and compared. The incidence and timing of MSSA/MRSA recolonization following decolonization with mupirocin will be determined. The incidence of nosocomial sepsis and invasive infections with any organisms will be determined and compared between the two groups. The incidence of mupirocin resistance in each group will be compared. The incidence of MSSA/MRSA colonization after discharge based on the outpatient screenings will be compared.

An independent study monitoring committee, composed of a pharmacist and an attending neonatologist (not the principal investigator), will meet after the first 30 patients are enrolled and periodically after the first review to ensure the safety of this study protocol for the duration of this study.

Rates of S. aureus colonization and infection during the study period will also be compared with historical rates from the Crouse Hospital NICU to ensure that there was not some other largely unanticipated change during the study period.

All study data will be compiled into an electronic database, which will be kept in a secure password-protected computer in the principal investigator's locked office on the ninth floor of Crouse Hospital. The study subjects' personal health information including name, date of birth, and medical record numbers will be used to identify subjects, and their study information will be part of their medical record. A copy of the data collection form and data analysis form will be submitted along with this protocol and application.

STATISTICAL METHODS, DATA ANALYSIS AND INTERPRETATION

Statistical analyses will include a descriptive phase to assess the frequencies of all variables and an analytic phase to evaluate the associations between methicillin-sensitivity or resistance status and the patient's gestational age, gender, birth weight, discharge diagnoses, discharge disposition, length of NICU stay, or presence/type of underlying condition, treatments, or clinical outcomes. Pearson's X2 test will be used to compare categorical variable counts/frequencies between the treatment and control groups. The two-sample t-test will be used for continuous variables with normal distribution to test differences between means. Appropriate alternatives, such as Wilcoxon rank sum, will be used if data violate t-test assumptions. The two-proportion z-test will be used to assess differences between two proportions. All hypothesis testing will be 2-tailed with a P ≤ 0.05 considered statistically significant. An analyst for statistical support has been involved with the study design, power analysis, and sample size calculation. She will remain involved throughout the study period and will assist with data analysis.

Neonatal MSSA/MRSA patient colonization days data from the Crouse Hospital NICU was used for sample size calculations. Approximately 12-15 new cases of MSSA- or MRSA-colonization occur each month, with a mean of 21.5 patient colonization days (standard deviation 20 days). A two-sample t-test with 95% confidence interval, power of 80, and hypothesized reduction of 40% (8 patient colonization days), suggests a sample size of 98 patients per group, or a total of approximately 200 patients in the study.

All study personnel, aside from the pharmacy staff who will randomize patients, will be blinded regarding patients' study group allocation until after discharge from the Crouse Hospital NICU. At time of discharge, the pharmacy will notify the principal investigator of each patient's study group allocation so that data analysis by treatment group can occur.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to Crouse Hospital NICU with MSSA/MRSA colonization that have parental consent for participation obtained within 2 days of their initial positive screen.

Exclusion Criteria:

* Any infant with an active or previous S. aureus infection at time of initial positive S. aureus colonization screen.
* Any infant with a condition thought to be fatal/irreversible (pulmonary hypoplasia, chromosomal/genetic syndromes, fatal cardiac anomalies).
* Any infant with a congenital condition that would prevent specimen collection or treatment application (cleft lip/palate, choanal atresia, abdominal wall defects, imperforate anus, etc.).
* Sufficient length of NICU admission will be necessary to adequately measure the primary outcome. Therefore, enrolled patients will only be included in data analysis if they remain in the NICU until after at least one subsequent MSSA/MRSA screening is performed following completion of their initial treatment course with either mupirocin or placebo.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Decolonization efficacy | Remaining length of NICU admission status post positive screening culture, approximately between 7 to 365 days
  Compare the number of S. aureus patient colonization days between treatment versus control group

SECONDARY OUTCOMES:
Trajectory of decolonization efficacy | Remaining length of NICU admission status post positive screening culture, approximately between 7 to 365 days
  Compare the proportions of persistently colonized, decolonized, and recolonized study subjects at each subsequent weekly screening interval in treatment versus control group
Incidence of recolonization | Remaining length of NICU admission status post positive screening culture, approximately between 7 to 365 days
  Determine the incidence and timing of recolonization with S. aureus following decolonization within the treatment group
Incidence of S. aureus infection | Remaining length of NICU admission status post positive screening culture, approximately between 7 to 365 days
  Determine and compare the incidence of nosocomial invasive S. aureus infection in treatment versus control group
Incidence of mupirocin-resistance | Remaining length of NICU admission status post positive screening culture, approximately between 7 to 365 days
  Determine the incidence of mupirocin-resistance in S. aureus isolates from treatment versus control group
Long-term decolonization efficacy | Within 2 months of discharge from NICU
  Determine and compare the incidence of S. aureus colonization between 1-2 months after discharge between treatment versus control group

CONTACTS AND LOCATIONS:
Overall Officials: Melissa U Nelson, MD, Principal Investigator — Crouse Hospital
Locations (1):
- Crouse Hospital - Neonatal Intensive Care Unit, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelson MU, Shaw J, Gross SJ. Randomized Placebo-Controlled Trial of Topical Mupirocin to Reduce Staphylococcus aureus Colonization in Infants in the Neonatal Intensive Care Unit. J Pediatr. 2021 Sep;236:70-77. doi: 10.1016/j.jpeds.2021.05.042. Epub 2021 May 21. PMID 34023342